CLINICAL TRIAL: NCT02428920
Title: Grenada Heart Project - Community Health Action to Encourage Healthy Behaviors
Acronym: GHP CHANGE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: St. George's University (Unknown)
Responsible Party: Principal Investigator, Valentin Fuster, Director, Mount Sinai Heart, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: GCO 12-2004
Record Dates: First submitted 2015-04-24; First posted 2015-04-29 (Estimated); Last update posted 2016-09-08 (Estimated); Status verified 2016-09

CONDITIONS: Health Behavior
Keywords: cardiovascular health; behavior change; community-based; prevention
MeSH Terms: conditions — Health Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Peer Groups (Experimental): Individuals in Intervention Group Arm will attend biweekly or monthly peer support groups (approximately 10 people per group) for evaluating changes and promoting mutual support. 12-month duration.
  Interventions: Behavioral: Peer Groups
- Control Arm (No Intervention): The control arm, will attend the initial educational group lectures at baseline assessment and will receive no intervention thereafter.

INTERVENTIONS:
Behavioral: Peer Groups — The intervention group arm will attend biweekly or monthly peer group meetings to discuss health successes and challenges.
  Arms: Peer Groups

SUMMARY:
The Grenada Heart Project (GHP) conducted an observational study within a randomly selected adult sample of Grenadians in 2008-2009. The aim of the study was to assess the clinical, biological and psychosocial determinants of the cardiovascular health in Grenada, in order to develop and implement a nationwide cardiovascular health promotion program.

The sample of 2,827 adults was randomly selected from the national electronic voter list. The main outcome measures were self-reported cardiovascular disease and behavioral risk factors, anthropometric measures, blood pressure (BP), point-of-care testing for glucose and lipids, and ankle-brachial index. Analysis of the data revealed prevalence rates of obesity, hypertension and diabetes significantly exceeding those seen in the U.S.

Since the completion of this assessment, an additional effort has contributed significantly to the current project. A parallel community health-promotion project was carried out in Cardona, Spain called the "Cardona Integral Fifty-Fifty" project with 80 subjects. The preliminary results of the Cardona study have a shown that peer motivation may significantly improve healthy behaviors and thus modify cardiovascular risk.

The GHP CHANGE community -based intervention aims to promote positive behaviors and focus more on what creates health, rather than what prevents sickness. It is built on the foundations of social support, assessing whether people going through similar challenges will support each other, work together to identify and address barriers to success, and motivate each other to move forward. In this program we test for the impact of promotion of healthy lifestyle behaviors through peer motivation on blood pressure, physical activity, eating behavior, weight, and smoking.

DETAILED DESCRIPTION:
This culturally-tailored intervention program will take place over a 12-month period in the following four regions on the island:

* St. David's Parish
* St. Andrew's Parish
* St. George's Parish
* St. John's/St. Mark's Parish (combined ) •The program will involve approximately 400 randomized participants (100 from each region). Participants, aged 18-70, from each parish will be divided into one of two groups: Intervention Group arm (peer support) or Control Group arm (individual study).

The investigators will identify study participants previously enrolled in the Grenada Heart Project, with at least one vascular risk factor, as defined by the Adult Treatment Panel III guidelines which include: elevated BP, increased blood glucose level, increased waist circumference, minimal reported physical activity, minimally reported fruit and vegetable intake, or current smoking habits. Given a 10% refusal rate and 10% failure rate in the run-in phase, 120 participants from each site will be invited randomly, from the high risk group, to recruit for participation in the study.

All eligible participants are invited to attend an informational half-day session, during which a general overview of the program is presented and participants have an opportunity to have any questions answered. During this session, eligible and interested individuals complete the written consent forms. Upon consenting, participants are informed of their randomization arm (education intervention or group intervention) and entered into a run-in phase. All participants receive a notebook, as well as certain health literate materials, provided by the American Heart Association. The educational materials will promote management of risk factors and the notebook will provide an avenue for recording of lifestyle behaviors, such as health goals, BP values, and eating habits.

•Participants enrolled in the run-in phase will complete the following assessments at three time points (baseline, 6-months, and 12-months):

* Anthropometric measurements
* GHP data collection form
* International physical activity questionnaire (iPAQ)
* Lifestyle Assessment [modified SF-36 questionnaire tailored to the Grenadian population]
* Point-of-care testing using an LDX analyzer (solely for the 12 month assessment).

The investigators have developed a "GHP Health outcomes Score" which captures a person's health profile on a 0-to-3 point scale related to smoking habits, overweight, sedentary lifestyle, and hypertension During the run-in phase, participants will attend a series of core lifestyle and risk factor education workshops related to motivation for change, nutrition (two sessions), smoking cessation, physical education and BP control. Only those participants who attend 4 of the 6 sessions will be eligible for randomization.

Eligible participants will be randomized to the intervention arm or to the control arm, stratified by parish. In the group intervention arm a group leader will be selected internally within the support groups, who will receive additional training from the research team in regards to group motivation and facilitation. Those randomized into the Intervention arm will be organized into peer groups of approximately 10 persons.

The specific aims of this study are:

Specific Aim 1: Hypothesis: Individuals will show an improvement of health-related behaviors through directed peer education groups (intervention group), compared to the individuals not receiving such peer support (control group).

Specific Aim 2: Hypothesis: Individuals will show an improvement in their quality of life through directed peer education groups (intervention group), compared to the individuals not receiving such peer support (control group).

Specific Aim 3: Hypothesis: Individuals will show an improvement in cardiovascular risk factors through directed peer education groups (intervention group), compared to the individuals not receiving such peer support (control group).

ELIGIBILITY:
Inclusion Criteria:

* Resident of Grenada
* One or more vascular risk factors:

  * Borderline to elevated blood pressure (defined as systolic blood pressure ≥120 mm Hg to SBP < 160 or diastolic blood pressure ≥ 80 and < 90 mm Hg)
  * Waist circumference of >40 inches for men and >35 inches for women
  * Smoking (active self-reported smoking, of any type of tobacco, at least daily)
  * Physical inactivity (reporting less than 120 min/week of activity)
  * Fasting glucose level > 100 mg/dl
  * Total Cholesterol >250 mg/dl, LDL > 130 mg/dl
  * Fruit/vegetable intake less than 2 servings daily

Exclusion Criteria:

* Unable/unwilling to provide consent
* Age of under 18 or more than 70 years old (inclusive) as of December 2012
* Inability of self-monitoring
* Pregnant women
* Morbidly ill with expectation of death within a year

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2014-07; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Composite GHP outcomes health score | baseline
  The GHP outcomes health score assimilates scores related to weight, diet, smoking, physical activity, blood pressure and quality of life.
Composite GHP outcomes health score | 6 months
  The GHP outcomes health score assimilates scores related to weight, diet, smoking, physical activity, blood pressure and quality of life.
Composite GHP outcomes health score | 12 months
  The GHP outcomes health score assimilates scores related to weight, diet, smoking, physical activity, blood pressure and quality of life.

SECONDARY OUTCOMES:
Change in blood pressure | baseline and 12 months
  Change in blood pressure at 12 months as compared to baseline
Change in body weight | baseline and 12 months
  Change in body weight at 12 months as compared to baseline
Change in behavior | baseline and 12 months
  Change in behavior as 12 months as compared to baseline

CONTACTS AND LOCATIONS:
Overall Officials: Valentin Fuster, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- St. George's University, Saint George's, Grenada

REFERENCES:
- [Derived] Latina J, Fernandez-Jimenez R, Bansilal S, Sartori S, Vedanthan R, Lewis M, Kofler C, Hunn M, Martin F, Bagiella E, Farkouh M, Fuster V. Grenada Heart Project-Community Health ActioN to EncouraGe healthy BEhaviors (GHP-CHANGE): A randomized control peer group-based lifestyle intervention. Am Heart J. 2020 Feb;220:20-28. doi: 10.1016/j.ahj.2019.08.022. Epub 2019 Sep 4. PMID 31765932